CLINICAL TRIAL: NCT02669745
Title: The Study of Molecular Risk Panels in Chinese Breast Cancer Patient Using Mammaprint, TargetPrint, BluePrint and Research Gene Panel Assays.
Brief Title: The Study of Molecular Risk Panels (70-gene Assay) in Chinese Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: P-0125
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Chinese
Keywords: Chinese women; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women of Chinese Descent: Females of Chinese descent, aged 18 year to 70 year, diagnosed with Stage 1 or Stage 2 (excluding those involving more than 3 lymph nodes) breast cancer.

SUMMARY:
This study is experimental and will prospectively assess the proportion of patients in the two (2) MammaPrint Risk categories in patients of Chinese descent.

DETAILED DESCRIPTION:
The incidence of breast cancer in Chinese women is lower than that of a Western population. Breast cancer is the most common cancer in Chinese women and the incidence is rising. Moreover there are more premenopausal women with breast cancer where the breast cancer incidence peaks in the forties and the postmenopausal rise in incidence is less commonly seen. As the genetic predisposition to breast cancer is increasingly understood, it has been suggested that the differences in breast cancer incidence in different ethnic populations is potentially due to interactions between lifestyle and genetic characteristics. To date, the use of Agendia's gene expression assays in Chinese women has not been studied. In this study, the feasibility of the gene-expression prognostic assays for risk assessment in this specific group will be assessed. Moreover, the specific molecular characteristics and potential biomarkers will be studied, focusing especially on the large group of premenopausal breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 year to 70 year,
* diagnosis of Stage I or Stage II (excluding those involving more than 3 lymph nodes) Breast Cancer
* Chinese descent

Exclusion Criteria:

* Stage II Breast Cancer with more than 3 positive lymph nodes

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women of Chinese Descent with Stage I or Stage II Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Comparing MammaPrint with Clinical Risk Assessment | 6 weeks
  The MammaPrint risk assessment outcomes will be compared with conventionally used risk assessments determined by clinical parameters, standard staging and IHC analysis (Adjuvant! Online) in a population of Chinese patients with breast cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided